CLINICAL TRIAL: NCT03209492
Title: Special Drug Use Surveillance of Leuplin PRO for Injection Kit 22.5 mg for "Prostate Cancer"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Leuprorelin-5002; JapicCTI-163213 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Results first posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Leuprorelin acetate: Usually, for adults, 22.5 mg of leuprorelin acetate is subcutaneously administered once every 24 weeks. Refer to the Precautions section of the package insert. Participants will receive interventions as part of routine medical care.
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: Leuprorelin acetate — Leuplin PRO for Injection Kit 22.5 mg
  Other Names: Leuplin PRO for Injection Kit 22.5 mg

SUMMARY:
The purpose of this study is to evaluate the safety in patients with prostate cancer receiving the drug in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this study is called Leuprorelin acetate (Leuplin PRO for Injection Kit 22.5 mg). Leuprorelin acetate is being tested to treat people who have prostate cancer.

This study will look at the safety in patients with prostate cancer receiving the drug in the routine clinical setting.

The study will enroll approximately 300 patients.

• Leuprorelin acetate

This multi-center trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants with prostate cancer will be included.

Exclusion Criteria:

* Participants with previous history of hypersensitivity to any of the ingredients of the drug or synthetic LH-RH or LH-RH derivatives

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of participants with a diagnosis of prostate cancer and received dose of Leuplin PRO for Injection Kit 22.5 mg/Leuprorelin acetate in the routine medical care.
Sampling Method: Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 61 investigative sites in Japan, from 01 April 2016 to 01 December 2017.
Pre-assignment Details: Participants with a historical diagnosis of prostate cancer were enrolled. Participants received interventions as part of routine medical care.
Groups:
- Leuprorelin Acetate 22.5 mg: Usually, for adults, 22.5 mg of Leuprorelin Acetate was subcutaneously administered once every 24 weeks. Refer to the Precautions section of the package insert. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Leuprorelin Acetate 22.5 mg
Started | 333
Completed | 328
Not Completed | 5
Not completed — Case Report Forms Uncollected | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the study.
Arm/Group | Leuprorelin Acetate 22.5 mg
Number analyzed (Participants) | 328
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.1 (6.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 328
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 328
Duration between Diagnosis of Prostate Cancer and Study Start [Mean (Standard Deviation); unit: Months] — Mean duration between the first diagnosis of prostate cancer and the start of the study was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Months
    number analyzed (Participants) | 323
    (all) | 53.15 (49.296)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Number of participants with each score of ECOG Performance Status at the study start was reported. Following are ECOG grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of self-care, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited self-care, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any self-care, totally confined to bed/chair.
  Participants
    0 | 243
    1 | 70
    2 | 6
    3 | 6
    4 | 3
Number of Participants who Had Treated with Adjuvant Therapy [Count of Participants; unit: Participants] | 36
Number of Participants with Localized Prostate Cancer [Count of Participants; unit: Participants] | 190
Number of Participants with Locally Advanced Prostate Cancer [Count of Participants; unit: Participants] | 45
Number of Participants with Metastatic Prostate Cancer [Count of Participants; unit: Participants] | 57
Number of Participants with Outpatient Care [Count of Participants; unit: Participants] | 328
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had No Predisposition to Hypersensitivity | 321
    Had Predisposition to Hypersensitivity | 5
    Unknown | 2
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Presence of Medical Complications | 109
    Had Presence of Medical Complications | 219
Medical History of Thromboembolism [Count of Participants; unit: Participants] — Number of participants with or without medical history of thromboembolism was reported.
  Participants
    Had No History of Thromboembolism | 293
    Had History of Thromboembolism | 33
    Unknown | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram per square meter (kg/m^2)
    number analyzed (Participants) | 250
    (all) | 23.49 (3.222)
Prior Treatment of LH-RH Agonists or Antagonist [Count of Participants; unit: Participants] — Number of participants who had or had not treated with LH-RH agonists or antagonist for prostate cancer was reported.
  Participants
    Not Treated with LH-RH Agonists or Antagonist | 31
    Treated with LH-RH Agonists or Antagonist | 297
Prior Treatment of Drugs for Prostate Cancer [Count of Participants; unit: Participants] — Number of participants who had or had not treated with drugs except LH-RH agonists or antagonist for prostate cancer was reported.
  Participants
    Not Treated with Drugs | 150
    Treated with Drugs | 178

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Events
Time Frame: Up to Week 24
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Leuprorelin Acetate 22.5 mg
Number analyzed (Participants) | 328
Percentage of Participants | 4.27

2. Secondary Outcome: Percentage of Participants Who Had One or More Adverse Reactions
Description: Adverse drug reaction refers to adverse events related to the administered drug.
Time Frame: Up to Week 24
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Leuprorelin Acetate 22.5 mg
Number analyzed (Participants) | 328
Percentage of Participants | 2.74

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Leuprorelin Acetate 22.5 mg
All-Cause Mortality (participants affected / at risk) | 4/328
Serious Adverse Events (participants affected / at risk) | 4/328
Other Adverse Events (participants affected / at risk) | 6/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin Acetate 22.5 mg (N=328)
Pneumonia (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Malaise (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin Acetate 22.5 mg (N=328)
Hot flush (Vascular disorders) | 3
Injection site induration (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT03209492/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03209492/SAP_001.pdf